CLINICAL TRIAL: NCT00074503
Title: Positron Emission Tomography Imaging of Incorporation of Docosahexaenoic Acid (DHA) From Plasma Into Human Brain
Brief Title: PET Imaging of DHA Metabolism
Status: Completed | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040058; 04-AA-0058
Record Dates: First submitted 2003-12-12; First posted 2003-12-15 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-07-13

CONDITIONS: Healthy
Keywords: Positron Emission Tomography; Phospholipids; Alcoholism; [11C]Docosahexaenoate; [150]Water; Brain; Fatty Acids; Blood Flow; Healthy
MeSH Terms: conditions — Alcoholism

SUMMARY:
This study will examine the use of positron emission tomography (PET) for measuring docosahexaenoic acid (DHA) absorption from the blood into the brain. DHA is a type of fatty acid found in fish and other seafood. It is involved in brain cell activity that underlies the ability to think, move, and respond to the outside world. When the amount of DHA in the brain is low, the brain may not work the same as if there were a normal amount of DHA. If PET can be used successfully to evaluate brain DHA metabolism, this method might be useful for future studies of alcoholism, since brain DHA levels are influenced by alcohol consumption.

Healthy normal volunteers between 18 and 65 years of age may be eligible for this study. Because study participants must stop taking any medications, including herbal preparations, individuals who require regular medication are excluded from this protocol. Participants will undergo the following tests and procedures:

* Psychological questionnaires concerning thoughts and behaviors.
* Nutritional status analysis: A dietitian will assess the subject's nutritional status through questionnaires and measurement of body fat. Body fat is measured using bioelectrical impedance analysis. This analysis uses a low, safe electric current to measure body composition, giving a reading of the percentage of fat in the body.
* Fat biopsy to measure the composition of fat tissue: An area on the upper half of the buttock will be numbed and a needle will be inserted to aspirate a sample of fat tissue for analysis.
* Blood drawing: Blood samples will be collected at the time of the fat biopsy and the PET scan (see below) to measure DHA and indicators that may influence DHA.
* Diet: 3 days before the fat biopsy and at least 3 days before the PET scan, subjects will consume a diet low in DHA and other omega-3 fats. This no seafood diet prohibits eating fish, shellfish, seaweed, seafood, health food products or supplemental vitamins, and foods containing canola or flaxseed oil. Caffeine-containing beverages are limited to one per day for 3 days before the study. Alcoholic beverages are prohibited for 2 weeks before the study. For 24 hours before the PET scan, subjects eat only standard meals that will be provided to them.
* Magnetic resonance imaging: A brain MRI scan will be done to fit the PET scan images onto a picture of the whole brain. During the scan, the subject lies on a table inside a narrow metal cylinder containing a strong magnetic field.
* PET scan: Before the PET scan, catheters (small plastic tubes) are inserted into an arm vein and into a wrist artery. The venous catheter is used for injecting a radioactive substance that will be detected by the scanner, and the arterial catheter is used for collecting blood samples during the scan. For the scan, the subject lies on a bed that slides into the doughnut-shaped scanner. A mask is placed to keep the head still. A transmission scan is done to see how much radiation the skull absorbs. Radioactive water (15O-water) is then injected into the blood, and the brain is scanned for about 10 minutes to measure brain blood flow. Then, radioactive DHA (11C-DHA) is injected, followed by about 1-1/2 hours of scanning to measure DHA absorption into the brain.

DETAILED DESCRIPTION:
Docosahexaenoic acid (DHA, 22:6 n-3) is an essential omega-3 fatty acid that is selectively concentrated in the brain. Epidemiologic studies suggest that DHA deficiency is related to affective disorders, while clinical studies suggest that DHA is efficacious in treating depression. DHA has also been shown to be an important second messenger involved in phospholipase A(2)-mediated signal transduction. Although animal studies have provided a wealth of knowledge about the role of DHA in neural function, no method exists of evaluating DHA content or metabolism in the living human brain. Our goal is to establish a quantitative method of examining brain DHA metabolism using PET in healthy humans and to measure regional DHA incorporation from plasma into the brain. Utilizing the data from the pilot phase with healthy volunteers, we will apply the method to study DHA metabolism in alcoholics. Since alcohol consumption depletes brain DHA, we hypothesize that compared to healthy volunteers; alcoholics will have a decreased rate of incorporation of DHA from plasma into brain. Utilizing the method we have established, we anticipate that we will find previously undetectable metabolic abnormalities in alcoholics. We may further find that such abnormalities are correlated with cognitive or behavioral function. Now that the pilot phase of the protocol has been completed, we are proceeding with the main phase of the protocol to study non-smoking chronic alcoholics.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 18-65 years.

EXCLUSION CRITERIA:

1. Any Axis I diagnosis, current or past.
2. History of any intravenous drug use, or a DSM IV diagnosis of drug use or alcohol abuse or dependence.
3. Recent use (within the past two weeks) of alcohol, or any period of extensive use, defined as an average of one standard drink per day over a twelve-month period.
4. Abnormal laboratory or diagnostic tests that might disturb the dependent measures of the study.
5. Inability to give a clinical history or informed consent.
6. Inability to follow dietary guidelines.
7. Serious medical problems requiring ongoing treatment (i.e., diabetes or hypertension).
8. Positive test for hepatitis C or human immunodeficiency virus (HIV).
9. Metallic foreign bodies lodged in the head or neck that would be affected by the MRI scanner magnet.
10. Head trauma resulting in a period of unconsciousness lasting longer than one hour.
11. History of central nervous system infection.
12. History of fetal alcohol syndrome or other neurodevelopment disorder.
13. History of seizures, other than in childhood and related to fever.
14. Nursing women, women with a positive pregnancy test or women of childbearing age who are not willing to use some form of birth control during the study.
15. Recent exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits of exposure.
16. Current use of cigarettes, cigars, or other form of tobacco, defined as ten cigarettes, two pipes or two cigars over the preceding month.
17. Current drug or medication use, or the use of any medication (i.e., Tylenol) for three days prior to PET.
18. Positive urine drug screen.
19. Psychotropic medication use (including benzodiazepines and illicit drugs) during the two weeks prior to the PET scan. The use of medication with a very long half life (i.e., Prozac) during the six weeks prior to the PET scan.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2003-12-12; Study Completion 2010-07-13

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bourre JM, Pascal G, Durand G, Masson M, Dumont O, Piciotti M. Alterations in the fatty acid composition of rat brain cells (neurons, astrocytes, and oligodendrocytes) and of subcellular fractions (myelin and synaptosomes) induced by a diet devoid of n-3 fatty acids. J Neurochem. 1984 Aug;43(2):342-8. doi: 10.1111/j.1471-4159.1984.tb00906.x. PMID 6736955
- [Background] Salem N Jr, Niebylski CD. The nervous system has an absolute molecular species requirement for proper function. Mol Membr Biol. 1995 Jan-Mar;12(1):131-4. doi: 10.3109/09687689509038508. PMID 7767372
- [Background] Bourre JM, Francois M, Youyou A, Dumont O, Piciotti M, Pascal G, Durand G. The effects of dietary alpha-linolenic acid on the composition of nerve membranes, enzymatic activity, amplitude of electrophysiological parameters, resistance to poisons and performance of learning tasks in rats. J Nutr. 1989 Dec;119(12):1880-92. doi: 10.1093/jn/119.12.1880. PMID 2576038